CLINICAL TRIAL: NCT07277465
Title: Role of the Microbiota in Obesity: Effect After Bariatric Surgery
Acronym: MICROOBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celia Bañuls (Other)
Responsible Party: Sponsor-Investigator, Celia Bañuls, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEIm: 8/21
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obese Patients With Bariatric Surgery
Keywords: obesity; gut microbiota; metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Bariatric Surgery; Anastomosis, Roux-en-Y

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bariatric surgery in patients with obesity (Experimental): Patients will undergo bariatric surgery if they meet the inclusion criteria and are willing to participate in the study.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery according to surgeon's assessment.
  Other Names: Roux en-Y bypass; sleeve gastrectomy; Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S)

SUMMARY:
Several studies have demonstrated that bariatric surgery is effective for inducing weight loss in obese patients. In addition, the effects of this surgery on multiple associated alterations are well known, including changes in the secretion and activity of hormones involved in appetite regulation, satiety, and energy expenditure, as well as alterations in the gut microbiota composition.

However, in cases of severe obesity, recent data have challenged the prevailing view, as bacterial species associated with low microbial richness (prior to surgery) appear to change only marginally after bariatric surgery, despite significant metabolic improvements.

Our objective is to examine whether gut microbiota and gastrointestinal peptides are further impaired in severe obesity and, additionally, to explore how the microbiota relates to metabolic profile or sex, as well as whether bariatric surgery may differentially correct obesity-related intestinal microbial features.

To this end, we propose a prospective, interventional, translational clinical study involving a cohort of 60 obese patients (BMI > 35 kg/m²) undergoing laparoscopic gastric bypass surgery. Patients will be grouped according to their degree of obesity to assess potential baseline differences and to evaluate the efficacy of the intervention. Furthermore, we will investigate whether these parameters differ according to metabolic profile or sex.

Body composition and nutritional status will be assessed, along with cardiovascular risk factors and comorbidities (hypertension, obstructive sleep apnea syndrome, dyslipidemia, type 2 diabetes mellitus, and insulin resistance). Gastrointestinal hormones (ghrelin, GIP, GLP-1, PYY, CCK, and leptin) will be measured in serum using Luminex XMAP technology. The content and diversity of the gut microbiota will be analyzed (16S rRNA amplicon sequencing and shotgun metagenomic sequencing using Illumina MiSeq technology) in stool samples collected before and 6-12 months after surgery. Additionally, individualized dietary follow-up and assessment of participants' quality of life will be conducted.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes mellitus (T2DM) continue to increase worldwide and are strongly associated with adverse metabolic and cardiovascular outcomes. Bariatric surgery, particularly laparoscopic gastric bypass (LGB), remains the most effective therapeutic strategy for substantial weight reduction, glycemic improvement, and favorable modulation of gastrointestinal hormones, bile acids, and gut microbiota. Nevertheless, the mechanisms explaining heterogeneous metabolic responses-especially in individuals with severe, morbid, or extreme obesity-remain insufficiently elucidated. In particular, gut microbial diversity, microbial gene richness, and related inflammatory pathways appear to contribute to metabolic health, yet their behavior in severe obesity and their evolution following bariatric surgery remain poorly characterized.

To address these gaps, the investigators designed a prospective, interventional, comparative, and translational clinical study including 60 obese individuals scheduled for bariatric surgery at a single tertiary hospital. Participants will be consecutively recruited according to strict inclusion and exclusion criteria and classified by degree of adiposity (severe, morbid, or extreme obesity), metabolic phenotype (metabolically healthy or metabolically abnormal obesity), and sex.

Prior to the surgical intervention, a structured dietary protocol will be implemented. Participants will receive an individualized hypocaloric diet tailored to nutritional requirements, with a macronutrient distribution of 55% carbohydrates, 30% fats, and 15% proteins. During the two weeks preceding surgery, a very low-calorie diet based on Optisource® sachets will be administered in three daily intakes. Postoperative dietary progression will follow standardized clinical guidelines, with close monitoring to support weight reduction and metabolic stabilization. Follow-up evaluations will occur at 1, 6, and 12 months after surgery.

All participants will undergo comprehensive baseline and longitudinal assessments, including: evaluation of nutritional status; anthropometric measurements; body composition and basal metabolism; cardiovascular risk factors; metabolic comorbidities; and exclusion of secondary causes of obesity. Analytical parameters will include fasting plasma glucose, lipid profile (triglycerides, HDL-cholesterol), blood pressure, markers of hepatic and renal function, and additional biochemical indices relevant to obesity and T2DM risk stratification. Gut microbiota profiling will be conducted to evaluate microbial composition, diversity, and gene richness. Gastrointestinal hormone analyses will quantify circulating incretins and appetite-regulating peptides, including GLP-1, PYY, and ghrelin, to explore their association with postoperative metabolic outcomes. Oxidative stress and inflammatory parameters will be also assessed in order to stratify cardiovascular risk before and after induced weight loss after bariatric surgery.

Statistical analyses will be performed using SPSS 17.0. Categorical variables will be summarized with frequency distributions and percentages. Quantitative variables will be described using mean, range, and standard deviation, with normality assessed via the Kolmogorov-Smirnov test. Between-group comparisons (sex, metabolic phenotype) will employ unpaired t-tests or Mann-Whitney U tests; comparisons across obesity categories will use ANOVA. Longitudinal changes following surgery will be evaluated with repeated measures ANOVA or paired t-tests. Correlations will be analyzed using Pearson or Spearman methods, and logistic regression models will be developed to identify predictive factors for specific metabolic responses.

This study aims to determine whether gut microbiota alterations are directly linked to metabolic abnormalities across obesity phenotypes and whether bariatric surgery elicits differential microbial and hormonal responses according to degree of adiposity and sex. It further explores whether gastrointestinal peptides and other peripheral biomarkers can refine obesity phenotyping and enhance individualized clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a body mass index (BMI) greater than 40 kg/m² (or > 35 kg/m² with minimum one obesity comorbidity).
* Aged between 18 and 65 years.
* Patients with a known duration of obesity exceeding five years, despite dietary interventions and farmacological treatment.

Exclusion Criteria:

* Due to the nature of the study, patients with acute or chronic inflammatory diseases, established hepatic or renal insufficiency (defined as transaminase levels ±2 SD from the mean and estimated glomerular filtration rate [CKD-EPI formula] >60), neoplasic diseases, or secondary causes of obesity (e.g., hypothyroidism, Cushing's syndrome) will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Analyze the changes in the diversity of the intestinal microbiota after bariatric surgery. | 5 years
  To assess the alpha-diversity of the intestinal microbiota, defined as the average diversity of species in an ecosystem, the Shannon index will be used. The results are interpreted as follows: values less than 2 are considered low in diversity and values greater than 3 are high in species diversity.
Assess differences in the diversity of the intestinal microbiota after bariatric surgery depending on the surgical procedure (Roux-en-Y gastric bypass vs sleeve gastrectomy vs SADI-S). | 5 years
  To assess the beta-diversity of the intestinal microbiota, defined as the average diversity of species in an ecosystem, the Bray-Curtis index will be used. The results are interpreted as follows: values less than 2 are considered low in diversity and values greater than 3 are high in species diversity.

SECONDARY OUTCOMES:
Evaluate the differences in the diversity of the intestinal microbiota depending on whether patients present metabolically healthy obesity (MHO) or metabolically unhealthy obesity (MUHO) before surgery | 5 years
  To asses the differences in alpha-diversity of the intestinal microbiota in both groups, it will be evaluated whether there are significant differences between the Shannon indices of the two groups. The classification of patients between MHO and MUHO will be carried out using the following criteria: MUHO will be considered when patients with obesity present ≥2 metabolic abnormalities, and MHO with ≤1 metabolic abnormalities; the following cardiovascular risk factors are considered metabolic abnormalities: elevated blood pressure (defined as either SBP ≥130 mm Hg, DBP ≥85 mm Hg, or treatment with antihypertensive medications), elevated triglycerides (as fasting triglyceride concentration ≥1.7 mmol/l), low HDL-C levels (defined as HDL-C <1.04 mmol/l, in men, <1.29 mmol/l/l in women, or treatment with lipid-lowering medications), dysglycemia (fasting plasma glucose 5.6 to 6.9 mmol/l, and/or and insulin resistance as HOMA-IR >3.8).
Evaluate significant changes in body fat mass percentage after bariatric surgery. | 3 years
  Percentage of body fat mass will be measured by bioelectrical impedance. It is considered to be high when ≥25% in men and ≥30% in women. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in high-sensitivity C-reactive protein (hs-CRP) as an inflammatory parameter after bariatric surgery. | 3 years
  Participants will be considered to have achieved an improvement in high-sensitivity C-reactive protein levels if they normalize its value (normality values defined between 0 and 1.69mg/dl).
Evaluate significant changes in C3 protein as an inflammatory parameter after bariatric surgery. | 3 years
  Participants will be considered to have achieved an improvement in C3 protein if they normalize its value (normality values defined between 81 and 157mg/dl).
Evaluate significant changes in interleukin 1-beta (IL-1B) levels as a pro-inflammatory molecule after bariatric surgery. | 3 years
  IL-1B levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in interleukin 6 (IL-6) levels as a pro-inflammatory molecule after bariatric surgery. | 3 years
  IL-6 levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in tumor necrosis factor alpha (TNF-alpha) levels as a pro-inflammatory molecule after bariatric surgery. | 3 years
  TNF-alpha levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in superoxide dismutase (SOD) levels after bariatric surgery. | 3 years
  Superoxide dismutase levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze the significant differences between metabolomic profile before and after bariatric surgery, and between different surgery procedures (Roux-en-Y gastric bypass vs. sleeve gastrectomy). | 3 years
  NMR spectra will be used to obtain spectra from serum samples from the cohort. In order to evaluate if there will be significant differences after the dietetic intervention, a PLS-DA model for discrimination between basal and post intervention levels will be performed. Scores plots will be calculated with a 95% confidence interval.
Evaluate if there is a significant reduction after bariatric surgery in total ROS levels. | 3 years
  Total ROS levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess if there is a significant reduction after bariatric surgery in glutathione levels. | 3 years
  Total glutathione levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant change after bariatric surgery in total free radicals levels. | 3 years
  Total free radicals will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant reduction after bariatric surgery in mitochondrial ROS production. | 3 years
  Mitochondrial ROS production will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate if there is a significant change after bariatric surgery in superoxide levels. | 3 years
  Superoxide content will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate if there is a significant improvement after bariatric surgery in mitochondrial membrane potential. | 3 years
  Mitochondrial membrane potential will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Identify and assess the differences in metabolic pathways of gut microbiota after bariatric surgery. | 5 years
  Genetic markers of inflammation and metabolic pathways will be analyzed from the faeces samples, in order to identify different clusters of these pathways and determine the potential functions of gut microbiota. For that purpose, transcriptome will be quantified with nanostring techology. The relative quantity of gene expression (fold change) of each gene will be calculated with the comparative 2-ΔΔCT method, and significant differences will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant reduction after the bariatric surgery in adipsin levels. | 3 years
  Adipsin levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in plasmatic resistin levels as an inflammatory parameter after surgical intervention. | 3 years
  Resistin levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant change after the bariatric surgery in leptin levels. | 3 years
  Leptin will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant reductions in Plasminogen activator inhibitor-1 (PAI-1) as an inflammatory parameter after the bariatric surgery. | 3 years
  PAI-1 levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess if there is a significant change after the bariatric surgery in ghrelin levels. | 3 years
  Ghrelin will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in serum Glucagon-like peptide-1 (GLP-1) levels after the bariatric surgery. | 3 years
  GLP-1 levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess if there is a significant improvement after bariatric surgery in peptide YY (PYY) levels. | 3 years
  PYY levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in serum gastric inhibitory polypeptide (GIP) levels after the bariatric surgery. | 3 years
  GIP levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze if there is a significant improvement after bariatric surgery in cholecystokinin (CCK) levels. | 3 years
  CCK levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nijhawan S, Richards W, O'Hea MF, Audia JP, Alvarez DF. Bariatric surgery rapidly improves mitochondrial respiration in morbidly obese patients. Surg Endosc. 2013 Dec;27(12):4569-73. doi: 10.1007/s00464-013-3125-y. Epub 2013 Aug 24. PMID 23982645
- [Background] Akalestou E, Miras AD, Rutter GA, le Roux CW. Mechanisms of Weight Loss After Obesity Surgery. Endocr Rev. 2022 Jan 12;43(1):19-34. doi: 10.1210/endrev/bnab022. PMID 34363458
- [Background] Ciobarca D, Catoi AF, Copaescu C, Miere D, Crisan G. Bariatric Surgery in Obesity: Effects on Gut Microbiota and Micronutrient Status. Nutrients. 2020 Jan 16;12(1):235. doi: 10.3390/nu12010235. PMID 31963247
- [Background] Cani PD, Van Hul M, Lefort C, Depommier C, Rastelli M, Everard A. Microbial regulation of organismal energy homeostasis. Nat Metab. 2019 Jan;1(1):34-46. doi: 10.1038/s42255-018-0017-4. Epub 2019 Jan 7. PMID 32694818
- [Background] Aron-Wisnewsky J, Prifti E, Belda E, Ichou F, Kayser BD, Dao MC, Verger EO, Hedjazi L, Bouillot JL, Chevallier JM, Pons N, Le Chatelier E, Levenez F, Ehrlich SD, Dore J, Zucker JD, Clement K. Major microbiota dysbiosis in severe obesity: fate after bariatric surgery. Gut. 2019 Jan;68(1):70-82. doi: 10.1136/gutjnl-2018-316103. Epub 2018 Jun 13. PMID 29899081
- [Background] Kootte RS, Levin E, Salojarvi J, Smits LP, Hartstra AV, Udayappan SD, Hermes G, Bouter KE, Koopen AM, Holst JJ, Knop FK, Blaak EE, Zhao J, Smidt H, Harms AC, Hankemeijer T, Bergman JJGHM, Romijn HA, Schaap FG, Olde Damink SWM, Ackermans MT, Dallinga-Thie GM, Zoetendal E, de Vos WM, Serlie MJ, Stroes ESG, Groen AK, Nieuwdorp M. Improvement of Insulin Sensitivity after Lean Donor Feces in Metabolic Syndrome Is Driven by Baseline Intestinal Microbiota Composition. Cell Metab. 2017 Oct 3;26(4):611-619.e6. doi: 10.1016/j.cmet.2017.09.008. PMID 28978426
- [Background] Sroka-Oleksiak A, Mlodzinska A, Bulanda M, Salamon D, Major P, Stanek M, Gosiewski T. Metagenomic Analysis of Duodenal Microbiota Reveals a Potential Biomarker of Dysbiosis in the Course of Obesity and Type 2 Diabetes: A Pilot Study. J Clin Med. 2020 Jan 29;9(2):369. doi: 10.3390/jcm9020369. PMID 32013181
- [Background] Amabebe E, Robert FO, Agbalalah T, Orubu ESF. Microbial dysbiosis-induced obesity: role of gut microbiota in homoeostasis of energy metabolism. Br J Nutr. 2020 May 28;123(10):1127-1137. doi: 10.1017/S0007114520000380. Epub 2020 Feb 3. PMID 32008579
- [Background] Bouter KE, van Raalte DH, Groen AK, Nieuwdorp M. Role of the Gut Microbiome in the Pathogenesis of Obesity and Obesity-Related Metabolic Dysfunction. Gastroenterology. 2017 May;152(7):1671-1678. doi: 10.1053/j.gastro.2016.12.048. Epub 2017 Feb 10. PMID 28192102
- [Background] Haluzik M, Kratochvilova H, Haluzikova D, Mraz M. Gut as an emerging organ for the treatment of diabetes: focus on mechanism of action of bariatric and endoscopic interventions. J Endocrinol. 2018 Apr;237(1):R1-R17. doi: 10.1530/JOE-17-0438. Epub 2018 Jan 29. PMID 29378901
- [Background] Murphy R, Clarke MG, Evennett NJ, John Robinson S, Lee Humphreys M, Hammodat H, Jones B, Kim DD, Cutfield R, Johnson MH, Plank LD, Booth MWC. Laparoscopic Sleeve Gastrectomy Versus Banded Roux-en-Y Gastric Bypass for Diabetes and Obesity: a Prospective Randomised Double-Blind Trial. Obes Surg. 2018 Feb;28(2):293-302. doi: 10.1007/s11695-017-2872-6. PMID 28840525
- [Background] Pareek M, Schauer PR, Kaplan LM, Leiter LA, Rubino F, Bhatt DL. Metabolic Surgery: Weight Loss, Diabetes, and Beyond. J Am Coll Cardiol. 2018 Feb 13;71(6):670-687. doi: 10.1016/j.jacc.2017.12.014. PMID 29420964